CLINICAL TRIAL: NCT02876029
Title: The Effect on Glucose Tolerance at a Second Meal Provided After Breakfast Meal Giving Late Increment in Postprandial Glycaemia
Brief Title: Food Design for Improved Day-long Glycaemic Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AFC-GPSecMeal
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Poor Glycemic Control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): White wheat bread
  Interventions: Other: Reference; Other: Test product
- Test product (Other): Pasta
  Interventions: Other: Reference; Other: Test product

INTERVENTIONS:
Other: Reference — the reference product used
  Other Names: WWB
Other: Test product — The test Product used
  Other Names: Pasta

SUMMARY:
The study focus is on the possible improvement in glucose tolerance at a second standardized meal that can be achieved when preceded by a test meal with a low GI and a high GP.

DETAILED DESCRIPTION:
A study in healthy subjects using spaghetti as the test breakfast and a white wheat bread as the reference. Glycaemia, insulinaemia, NEFA, TG and subjective appetite are studied up to the time of the lunch meal that is served 4h after breakfast. After lunch the blood sampling continues for 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-25

Exclusion Criteria:

* Smoker, Diabetes, Gluten intolerance, vegetarian

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Glucose | 0-6 h

SECONDARY OUTCOMES:
Non-esterified fatty acids (NEFA) | 0-6 h
Triglycerides (TG) | 0-6 h
Appetite rating (Visual Analogue Scale) | 0-6 h
Insulin | 0-6 h

CONTACTS AND LOCATIONS:
Overall Officials: Elin Östman, Ass prof, Study Director — Food for Health Science Centre (Medicon Village) - Lund University

IPD SHARING:
Plan to Share IPD: No